CLINICAL TRIAL: NCT05358899
Title: The Effect and Safety of Accelerated Continuous Theta-burst Stimulation on Metabolic Dysfunction in People With Schizophrenia
Brief Title: Accelerated cTBS on Metabolic Dysfunction in People With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: wu2022acTBS
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Schizophrenia; Metabolic Disturbance; Eating Behavior; Transcranial Magnetic Stimulation
Keywords: schizophrenia; metabolic disturbance; cTBS; Event related potentials
MeSH Terms: conditions — Schizophrenia; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Quadro-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care provider, investigator, and outcome assessor will be blind to the intervention except the treatment provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real stimulation (Experimental): Participants in the real stimulation group will receive accelerated cTBS with 1800 stimulation per session for 10 consecutive days, 5 sessions per day with a gap at least one hour, 50 sessions in total. The stimulation will be conducted at left M1 area.
  Interventions: Device: accelerated theta burst stimulation
- Sham stimulation (Sham Comparator): Participants in the sham stimulation group will receive the stimulation with coil vertical to the surface with other settings same as the real stimulation group.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: accelerated theta burst stimulation — cTBS was administered at 80% of each participant's M1 area in a burst-firing pattern (3 pulses at 50 Hz) with a repetition frequency of 5 Hz (200 ms intervals). During each session, participants received 1800 pulses (120 s).
  Arms: Real stimulation
Device: Sham stimulation — Similar process with the accelerated theta burst stimulation with the coil 90 degrees tilted to the surface of the scalp, which could produce identical sound and vibration while avoiding real magnetic stimulation.
  Arms: Sham stimulation

SUMMARY:
cTBS is a promising novel intervention, which has strong potential on moderating disease syndrome. However, the most effective pattern of the cTBS is still under debate. Therefore, the investigators designed this randomized controlled clinical trial to evaluate the efficacy and safety of accelerated cTBS, with 1800 stimulation per session, on intervention to metabolic side effects in individuals with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia in accordance with DSM-5
* BMI over 24
* Accepting antipsychotics stable treatment for more then 2 months

Exclusion Criteria:

* Diagnosed with other mental disease in accordance with DSM-5
* Comorbid with other severe physiological disease
* Used antipsychotic, antidepressants, mood stabilizer, or other psychoactive substances before
* Drug or alcohol abuse
* Pregnant or lactating Contraindication to rTMS

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of body weight | from baseline to 6 weeks
  the change of participants weight
Change of body mass index | from baseline to 6 weeks
  the change of participants BMI

SECONDARY OUTCOMES:
Positive and Negative syndrome rating scale | from baseline to 6 weeks
  Positive and Negative syndrome rating scale, from 30-210, higher score means worse symptoms.
Three Factor Eating Questionnaire | from baseline to 6 weeks
  three domain regarding eating behavior, from 0-51, higher score means better.
Barrat impulsiveness scale | from baseline to 6 weeks
  four domains regarding impulsiveness, from 26-104 higher score means higher impulse.
Self-Control Scale | from baseline to 6 weeks
  five domains regarding self control ability, from 36-180 higher score means better self control.
Food picture stimulation Event-related potentials | from baseline to 6 weeks
  Several components of event-related potentials were analyzed regarding various cognitive processes. The data were analyzed using previously widely used pipelines to extract the characters of ERP components, for example, P3 and LPP, and compare its difference within groups and between groups through time. ERP analysis will be conducted using EEGLAB and FieldTrip in MATLAB, and statistic analysis will be conducted using R studio and SPSS.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
The data will be provided for scientific study only with the permission of the principle investigator.